CLINICAL TRIAL: NCT00289406
Title: An 8 Weeks, Multi-Center, Randomized, Double Blinded, Comparative Phase 3 Clinical Trial to Assess the Efficacy and Safety of S-Amlodipine Gentisate Compared to Amlodipine Besylate in Patients With Mild-to-Moderate Hypertension
Brief Title: Efficacy and Safety Study of S-Amlodipine Gentisate Compared to Amlodipine Besylate to Treat Mild-to-Moderate Hypertension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: SK Chemicals Co., Ltd. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SK310_III_2006
Record Dates: First submitted 2006-02-07; First posted 2006-02-09 (Estimated); Last update posted 2007-03-06 (Estimated); Status verified 2006-09

CONDITIONS: Hypertension
Keywords: hypertension
MeSH Terms: conditions — Hypertension | interventions — Amlodipine

INTERVENTIONS:
Drug: S-amlodipine gentisate
Drug: Amlodipine besylate

SUMMARY:
The goal of this study is to compare the antihypertensive effect and tolerability of S-amlodipine gentisate with those of amlodipine besylate in patients with mild to moderate hypertension.

ELIGIBILITY:
Inclusion Criteria:

* patients are required to have a mean cuff sitting diastolic blood pressure of ≥90 and ≤109 mmHg after successful completion of the 2-week placebo run-in period

Exclusion Criteria:

* any serious disorder that could limit the ability of the patient to participate in the study
* significant cardiovascular disease (angina, myocardial infarction, cerebrovascular disease, or significant arrhythmia in the preceding 6 months)
* uncontrolled diabetes mellitus (serum glucose level ≥140 mg/dl)
* insulin dependent diabetes mellitus (type I)
* secondary hypertension

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110
Dates: Start 2006-01; Study Completion 2006-02

PRIMARY OUTCOMES:
The difference in mean changes from baseline in through sitting diastolic blood pressure after 8 weeks of treatment

SECONDARY OUTCOMES:
Mean changes in sitting systolic blood pressure; response rate (defined as the proportion of patients whose sDBP was ≤90mmHg or whose sDBP had decreased from baseline by ≥10 mmHg); changes in triglyceride and total cholesterol level of blood sample

CONTACTS AND LOCATIONS:
Overall Officials: SK Chemicals Investigational Site Seoul, Professor, Principal Investigator — SK Chemicals Investigational Site
Locations (1):
- SKChemicals, Seoul, South Korea